CLINICAL TRIAL: NCT06277102
Title: Effects of Music on Acute Postoperative Pain Intensity and Mobility After Fragility Hip Fracture: A Randomized Controlled Trial
Brief Title: Effects of Music on Acute Postoperative Pain Intensity and Mobility After Fragility Hip Fracture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Lau Kwan Yiu Jeffrey, Advanced Practice Nurse, Hospital Authority, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Music pain FHF
Record Dates: First submitted 2024-02-08; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Hip Fractures
Keywords: pain control; music; fragility hip fracture
MeSH Terms: conditions — Hip Fractures; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music (Experimental): Music listening at postoperative day 1 and 2, 1 session per day, 20 minutes per session.
  Interventions: Other: music listening
- Control (No Intervention): Standard of care

INTERVENTIONS:
Other: music listening — Music listening at postoperative day 1 and 2, 1 session per day, 20 minutes per session.
  Arms: Music

SUMMARY:
Music has been proven to be beneficial in postoperative care by reducing pain. The effects of music listening to reduce pain postoperatively are well studied among cases undergoing elective orthopaedic surgery. No study has been conducted focusing on pain control among cases with fragility hip fractures in an acute ward setting with non-schedule non-elective orthopaedic operation.

In Queen Elizabeth Hospital a standardized analgesic protocol is used for all fragility hip fracture cases unless contraindicated, a suboptimal post-operative pain control is not uncommonly seen. Stepping up analgesics is usually a concern in the elderly with a higher rate of side effects, a safe and simple non-pharmacological intervention for pain control is therefore needed.

The aim of this study is to study the effectiveness of incorporating music on pain intensity and mobility with the standard postoperative rehabilitation care of fragility hip fracture in Queen Elizabeth Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Emergency admitted to QEH/G9 due to fragility hip fracture (#NOF or # TOF) within the study period
2. Plan for surgical intervention
3. Able to provide written informed consent
4. Able to communicate in Cantonese/ Putonghua/ English

Exclusion Criteria:

1. History of dementia
2. Acute delirium upon admission
3. Disorientated to time, person or place
4. Concurrent fracture at other sites
5. Utilization of other analgesics on top of pain protocol
6. Appreciable deficits in hearing or vision
7. Hemodynamically unstable
8. Plan for neurolysis/ nerve block as definite treatment or opt for conservative treatment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity measured by 11-point pain intensity numerical rating scale after music listening in postoperative Day 1 - 2 among subjects with fragility hip fracture | postoperative day 1 and 2

SECONDARY OUTCOMES:
Modified functional ambulatory classification (MFAC) in postoperative Day 3 among subjects with fragility hip fracture | postoperative day 3
New mobility score (NMS) in postoperative Day 3 among subjects with fragility hip fracture | postoperative day 3

CONTACTS AND LOCATIONS:
Locations (1):
- Ward G9, Queen Elizabeth Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No